CLINICAL TRIAL: NCT07228351
Title: Comparison of the Effects of Vaginal Cuff Closure Techniques on Vaginal Length and Sexual Function in Laparoscopic Hysterectomy
Brief Title: Comparison of the Effects of Vaginal Cuff Closure Sexual Function in Laparoscopic Hysterectomy
Status: Available | Type: Expanded Access
Sponsor: Acibadem Kent Hospital (Other)
Responsible Party: Principal Investigator, merve ecem albayrak, Medical doctor, Acibadem Kent Hospital
Other Study IDs: AcibademKentH
Record Dates: First submitted 2025-11-10; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Uterus Absent
Keywords: hysterectomy; laparoscopy; suturation
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Behavioral: The effect of the vaginal cuff closure technique on women's sexual life and urogenital functions — The Arizona Sexual Experiences Scale is a 6-point Likert-type scale consisting of 5 questions. The lowest possible score is 5, and the highest is 30. Scores of 11 or more are considered sexual dysfunction.
Device: ultrasound — Vaginal length measurement accompanied by ultrasound

SUMMARY:
Aim: Laparoscopic hysterectomy is the vaginal removal of the uterus with the help of laparoscopy. After the uterus is removed after hysterectomy, vaginal length is shortened by cuff suturing, resulting in conditions such as dyspareunia and sexual dysfunction . Hysterectomy may also affect women physically and psychologically, as well as causing changes in sexual functions . In patients planned to undergo hysterectomy; Changes that may occur in sexual functions cause serious concerns during the preoperative period. However, physicians often miss these important points and do not discuss these issues adequately with patients. In this study; We aimed to compare the effects of vaginal cuff closure techniques in laparoscopic hysterectomy on vaginal length and women's sexual life. We used the Arizona Sexual Experience Scale to assess women's sexual life.

DETAILED DESCRIPTION:
Hysterectomy, defined as the surgical removal of the uterus, is one of the most commonly performed gynecological operations worldwide. Indications for hysterectomy, which is frequently performed on women of reproductive age and menopause, are emphasized in the literature as including pelvic masses (uterine myomas), abnormal bleeding (menorrhagia, menometrorrhagia, dysfunctional uterine bleeding), ovarian cysts, endometriosis, pelvic pain, pelvic prolapse, and urinary incontinence. Currently, there are many approaches to hysterectomy. The uterus can be removed abdominally, vaginally, laparoscopically, or robotically. Due to the advantages of minimally invasive surgery, laparoscopic and robotic hysterectomies are on the rise, while the rate of vaginal and abdominal hysterectomies is decreasing. Laparoscopic hysterectomy is the vaginal removal of the uterus using laparoscopy. Advantages include rapid postoperative recovery, short hospital stay, reduced need for analgesia, and improved visualization of the pelvic organs. Hysterectomy can lead to bleeding, infection, thromboembolic events, and gastrointestinal and urinary complications. Due to the removal of the uterus after hysterectomy, vaginal length shortens, leading to conditions such as dyspareunia and sexual dysfunction. Hysterectomy can also affect women physically and psychologically, as well as alter sexual function. Sexual function after hysterectomy can be affected by physiological factors (reduced tissue quality, neural stimulation, and pelvic blood flow due to anatomical changes in pelvic tissue), hormonal factors (reduced ovarian blood flow or decreased estrogen and progesterone levels due to the removal of the ovaries along with hysterectomy), psychological factors (depression, altered body image, and perception of femininity), and factors related to the hysterectomy technique. There are conflicting opinions regarding the effect of the uterus on sexual function. Some authors suggest that uterine contractions play an important role in the orgasmic phase, while others suggest that hysterectomy causes vaginal shortening or damage to autonomic nerve endings in the cervicovaginal area, leading to sexual dysfunction. The causal relationship between hysterectomy and decreased sexual function has been linked to shortened vaginal length and the emergence of postoperative dyspareunia. This is influenced by the vaginal cuff closure techniques used during hysterectomy.

Research on the relationship between hysterectomy and postoperative urinary incontinence or urogenital complaints has yielded mixed results. Studies report varying effects of hysterectomy on urinary incontinence. However, it is unclear whether postoperative urinary incontinence is due to the hysterectomy itself, influenced by the technique, or due to preoperative factors. The possibility of deterioration in sexual function and urinary dysfunction in patients undergoing hysterectomy raises serious concerns during the preoperative period. However, physicians often overlook these important points and fail to adequately discuss them with patients. In this study, we aimed to investigate the effects of the vaginal cuff closure technique in laparoscopic hysterectomy on women's sexual life and urogenital functions. We used the Arizona Sexual Experiences Scale and vaginal length measurement to assess women's sexual life, and the Urogenital Distress Inventory to assess urogenital functions. Patients who underwent laparoscopic hysterectomy at the Obstetrics and Gynecology Department of Abant İzzet Baysal University Faculty of Medicine will be included in this study. Patients who underwent total laparoscopic hysterectomy will be divided into two groups based on the vaginal cuff closure technique: laparoscopic and vaginal. Patients will be recorded and evaluated based on their age, gender, parity, body mass index, presenting complaints, ultrasonography findings, probe curettage results, Pap smear results, surgical indications, current chronic diseases, and past surgical history. Data obtained in the study will be analyzed using SPSS. During total laparoscopic hysterectomy, vaginal cuff closure techniques will be used to divide the patients into two groups: laparoscopic and vaginal closure.

ELIGIBILITY:
Inclusion Criteria:

* Perimenopausal period
* Having undergone surgery for benign gynecological indications
* Complete and accurate patient registration information.
* Volunteering to participate in the study.

Exclusion Criteria:

* Uterus size greater than 14 weeks' gestation
* Pelvic organ prolapse in the preoperative period
* Urinary incontinence in the preoperative period
* Cases with intraoperative complications
* Having undergone another concurrent surgery (urinary incontinence surgery, bowel surgery, etc.)
* History of endometriosis
* History of pelvic inflammatory disease

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- İzmir Kent Acibadem Hospital, Izmir, Turkey (Türkiye)

REFERENCES:
- [Result] Turner LC, Shepherd JP, Wang L, Bunker CH, Lowder JL. Hysterectomy surgery trends: a more accurate depiction of the last decade? Am J Obstet Gynecol. 2013 Apr;208(4):277.e1-7. doi: 10.1016/j.ajog.2013.01.022. Epub 2013 Jan 17. PMID 23333543

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-01): https://cdn.clinicaltrials.gov/large-docs/51/NCT07228351/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-01): https://cdn.clinicaltrials.gov/large-docs/51/NCT07228351/ICF_001.pdf